CLINICAL TRIAL: NCT06763744
Title: SMart Angioplasty Research Team- Genotype-Guided Abbreviated DUal AntIplatelet Therapy Versus Un-Guided De-escalation Therapy in Patients With Acute Coronary SyndromE and High Bleeding Risk (SMART-GUIDE-HBR)
Brief Title: Genotype-Guided Abbreviated DAPT Versus Un-Guided De-escalation Therapy in Patients With ACS and HBR
Acronym: GUIDE-HBR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUIDE-HBR
Record Dates: First submitted 2025-01-01; First posted 2025-01-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Coronary Syndrome (ACS) Undergoing Percutaneous Coronary Intervention (PCI); High Bleeding Risk
Keywords: CYP2C19 Genotype; Acute coronary syndrome; De-escalation therapy; P2Y12 inhibitor monotherapy; High bleeding risk
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, two-arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genotype-guided abbreviated DAPT (Active Comparator): Rapid (CYP2C19*1/*17 or *17/*17) or normal metabolizers (CYP2C19*1/*1) for clopidogrel will receive clopidogrel monotherapy and intermediate or poor metabolizers will receive potent P2Y12 inhibitor (prasugrel or ticagrelor) monotherapy (patients carrying a CYP2C19*2 or *3 alleles) after 1 month of potent P2Y12 inhibitor based DAPT.
  Interventions: Drug: P2Y12 antagonist monotherapy
- Un-guided de-escalation of DAPT (Active Comparator): A potent P2Y12 inhibitor is changed to clopidogrel 1 month after PCI, and aspirin is maintained.
  Interventions: Drug: clopidogrel + aspirin

INTERVENTIONS:
Drug: P2Y12 antagonist monotherapy — CYP2C19 genetic testing is performed before discharge after stent insertion. Depending on the test results, rapid (CYP2C19*1/*17 or *17/*17) or normal (CYP2C19*1/*1) metabolizers are treated with clopidogrel monotherapy, and intermediate or poor metabolizers (with CYP2C19*2 or *3 alleles) are treated with potent P2Y12 inhibitors (prasugrel or ticagrelor) monotherapy.
  Arms: Genotype-guided abbreviated DAPT
Drug: clopidogrel + aspirin — In this group, a potent P2Y12 inhibitor was changed to clopidogrel (un-guided) 1 month after PCI with maintenance of co-prescription of aspirin (DAPT).
  Arms: Un-guided de-escalation of DAPT

SUMMARY:
The aim of this study is to assess the safety and efficacy of the CYP2C19 genotype-guided abbreviated dual antiplatelet therapy (DAPT) strategy versus the un-guided stepwise intensity de-escalation of DAPT strategy in patients with acute coronary syndrome (ACS) and high bleeding risk (HBR) undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Current guidelines recommend reducing the duration of dual antiplatelet therapy (abbreviated DAPT) or de-escalating P2Y12 inhibitor intensity (de-escalation therapy) in patients at risk of major bleeding, even in patients with acute coronary syndromes. A network meta-analysis that indirectly compared these two strategies found that abbreviated dual antiplatelet therapy reduced major bleeding compared with de-escalated dual antiplatelet therapy.

Unlike prasugrel and ticagrelor, which are potent P2Y12 inhibitors, clopidogrel is activated in the liver via the cytochrome P450 2C19 (CYP2C19) metabolic pathway to exert its antiplatelet effects. Its use as monotherapy requires caution, given that CYP2C19 genotypes that may be resistant to clopidogrel are more prevalent in Asian populations than in Western populations.

Therefore, this study aimed to compare the clinical outcomes and confirm the efficacy and safety of an abbreviated dual antiplatelet therapy (Abbreviated DAPT, P2Y12 inhibitor monotherapy) strategy based on CYP2C19 genetic testing and a step-down DAPT strategy (De-escalation therapy) after 1 month of maintenance potent P2Y12 inhibitor-based dual antiplatelet therapy in patients at HBR who underwent PCI for ACS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 19 years of age
* Patients who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily.
* Patients presenting with ACS (ST-elevation myocardial infarction [STEMI] or non-ST-elevation [NSTE] ACS).
* Patients with at least one lesion with equal or greater than 50% diameter stenosis requiring treatment with drug-eluting stents in native coronary artery or graft.
* Patients with high bleeding risk (by ARC-HBR definition or PRECISE-DAPT score 25 or more)

Exclusion Criteria:

* Patients unable to provide consent.
* Patients who need chronic anti-coagulation therapy.
* Patients suffering from cardiogenic shock or cardiac arrest
* Patients with known intolerance to aspirin, all P2Y12 inhibitors, or components of drug-eluting stents.
* Clinically significant out of range values for platelet count (< 50,000/mm3) or hemoglobin (<8 g/dL) at screening
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Pregnant or lactating women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Major or clinically relevant non-major bleeding | 6 months after PCI
  Bleeding Academic Research Consortium type 2, 3, or 5

SECONDARY OUTCOMES:
Major bleeding | 6 months after PCI
  BARC type 3 or 5
Clinically relevant non-major bleeding | 6 months after PCI
  BARC type 2
Net adverse clinical event | 6 months after PCI
  A composite of all-cause death, MI, stroke, stent thrombosis, and major bleeding
Major adverse cardiac and cerebrovascular event | 6 months after PCI
  A composite of all-cause death, MI, stent thrombosis, or stroke
All-cause death | 6 months after PCI
  Death from any causes
Cardiovascular death | 6 months after PCI
  Death from cardiovascular causes
MI | 6 months after PCI
Stent thrombosis | 6 months after PCI
  Definite or probable, defined by ARC
Stroke | 6 months after PCI
Repeat revascularization | 6 months after PCI
Target vessel revascularization | 6 months after PCI
Target lesion revascularization | 6 months after PCI
A composite of cardiovascular death, MI, stent thrombosis, or stroke | 6 months after PCI
A composite of cardiovascular death, MI, stent thrombosis, stroke, or repeat revascularization | 6 months after PCI
Total medical cost | 1 year after PCI
Major or clinically relevant non-major bleeding | 1 year after PCI
Major bleeding | 1 year after PCI
Clinically relevant non-major bleeding | 1 year after PCI
Net adverse clinical event | 1 year after PCI
  A composite of all-cause death, MI, stent thrombosis, stroke, and major bleeding
Major adverse cardiac and cerebrovascular event | 1 year after PCI
  A composite of all-cause death, MI, stent thrombosis, or stroke
All-cause death | 1 year after PCI
Cardiovascular death | 1 year after PCI
MI | 1 year after PCI
Stent thrombosis | 1 year after PCI
Stroke | 1 year after PCI
Repeat revascularization | 1 year after PCI
Target vessel revascularization | 1 year after PCI
Target lesion revascularization | 1 year after PCI
A composite of cardiovascular death, MI, stent thrombosis, or stroke | 1 year after PCI
A composite of cardiovascular death, MI, stent thrombosis, stroke, or repeat revascularization | 1 year after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided